CLINICAL TRIAL: NCT00666185
Title: A Phase 3, Randomized, Double-Blind, Comparative Trial of Micafungin Versus Fluconazole for the Treatment of Esophageal Candidiasis
Brief Title: Comparative Trial of Micafungin Versus Fluconazole for Treating Esophageal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-7-005
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Candidiasis, Oral
Keywords: Micafungin; Esophageal Candidiasis; Fluconazole
MeSH Terms: conditions — Candidiasis, Oral | interventions — Micafungin; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Micafungin
- 2 (Active Comparator)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: Mycamine; FK463
  Arms: 1
Drug: Fluconazole — IV
  Other Names: Diflucan
  Arms: 2

SUMMARY:
To determine the efficacy and safety of IV Micafungin versus IV Fluconazole in the treatment of patients with Esophageal Candidiasis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of esophageal candidiasis confirmed by endoscopy
* Negative pregnancy test in females of childbearing potential

Exclusion Criteria:

* Pregnant or nursing
* Evidence of liver disease
* Presence of another active opportunistic fungal infection and/or receiving acute systemic therapy for an opportunistic fungal infection
* Concomitant esophagitis caused by herpes simplex virus or cytomegalovirus
* Receipt of an oral or topical antifungal agent within 48 hours or a systemic agent within 72 hours of first dose of study drug
* Non-responsive to therapy in any prior systemic antifungal clinical trail
* History of > 2 episodes of esophageal candidiasis requiring systemic antifungal therapy
* History of anaphylaxis attributed to azole compounds or echinocandin class of antifungals

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2003-08; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Endoscopic cure rate, defined as a mucosal grade of zero at the end of the therapy | End of Therapy

SECONDARY OUTCOMES:
Clinical response at end of therapy of cleared or improved | End of Therapy
Mucosal response at end of therapy of cleared or improved | End of Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Director — Astellas Pharma US, Inc.
Locations (37):
- Brazil (16):
  - Abadia Uberaba
  - Barretos
  - 5 Sites, Belo Horizonte
  - Boqueirao - Santos
  - 2 Sites, Campinas
  - 2 Sites, Curitiba
  - Goiânia
  - Maruipe Victoria
  - Nova Iguaçu
  - Parquelandia - Fortaleza
  - Porto Alegre
  - Quinta - Natal
  - 4 Sites, Rio de Janeiro
  - 2 Sites, Salvador
  - São José do Rio Preto
  - 8 Sites, São Paulo
- 4 Sites, Lima, Peru
- South Africa (20):
  - Arcadia-Pretoria
  - Bellville - Cape Town
  - 2 Sites, Bloemfontein
  - Brits
  - Cape Town
  - Centurion
  - Dundee
  - 2 Sites, Durban
  - Hatfield - Pretoria
  - Johannesburg
  - Olifantsfontein
  - Paarl
  - 2 Sites, Port Elizabeth
  - Potchefstroom
  - 3 Sites, Pretoria
  - Pretoria West
  - Reiger Park
  - Richards Bay
  - Somerset West
  - Westdene - Bloemfontein

REFERENCES:
- [Background] de Wet NT, Bester AJ, Viljoen JJ, Filho F, Suleiman JM, Ticona E, Llanos EA, Fisco C, Lau W, Buell D. A randomized, double blind, comparative trial of micafungin (FK463) vs. fluconazole for the treatment of oesophageal candidiasis. Aliment Pharmacol Ther. 2005 Apr 1;21(7):899-907. doi: 10.1111/j.1365-2036.2005.02427.x. PMID 15801925
- [Derived] Andes DR, Reynolds DK, Van Wart SA, Lepak AJ, Kovanda LL, Bhavnani SM. Clinical pharmacodynamic index identification for micafungin in esophageal candidiasis: dosing strategy optimization. Antimicrob Agents Chemother. 2013 Nov;57(11):5714-6. doi: 10.1128/AAC.01057-13. Epub 2013 Aug 19. PMID 23959319